CLINICAL TRIAL: NCT06271096
Title: Intramuscular Midazolam Versus Intravenous Diazepam for Acute Seizure in Children
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Arooj Khan (Other)
Responsible Party: Sponsor-Investigator, Arooj Khan, Assistant Professor Muhammad Kashif, Khyber Teaching Hospital
Organization: Khyber Teaching Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 638/ADR/KMC
Record Dates: First submitted 2024-02-07; First posted 2024-02-21 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Seizures
MeSH Terms: conditions — Seizures

STUDY DESIGN:
Intervention Model Description: This study was a randomized controlled trial carried out between November 2019 to November 2022 in the Pediatric department of Khyber Teaching Hospital. A total of 150 children who presented to the emergency department with seizures were enrolled in this study via consecutive sampling. This study was approved by the Ethical Review
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A IM-Midazolam (Experimental): Group A received IM midazolam at a dose of 0.2 mg/kg gently injected into the vastus lateralis muscle
  Interventions: Drug: Intra muscular Midazolam
- Group B IV Diazepam (Experimental): Patients in group B were cannulated in the dorsum of the hand or foot, or the great saphenous vein at the ankle first and then administered diazepam at a dose of 0.2mg/kg
  Interventions: Drug: Intravascular Diazepam

INTERVENTIONS:
Drug: Intra muscular Midazolam — ROUTE OF ADMINISTRATION AND DRUG EFFICACY COMPARED
  Arms: Group A IM-Midazolam
Drug: Intravascular Diazepam — ROUTE OF ADMINISTRATION AND DRUG EFFICACY COMPARED
  Arms: Group B IV Diazepam

SUMMARY:
IM-midazolam in acute seizures, whenever IV cannulation is not possible. It is easy to administer and can be used in prehospital settings as IV cannulation requires experience, especially in pediatric age group. Moreover, the transit time to the hospital can be prolonged in our areas which can delay the treatment if intravenous cannulation is considered. More studies are required to assess the feasibility of administering IM-midazolam in a prehospital setting to control acute seizures

DETAILED DESCRIPTION:
A seizure or convulsion is a time-limited, paroxysmal, change in motor activity and or behavior that results from electrical activity in the brain that is abnormal.1 The emergency department of a hospital is usually the place where children with seizures receive first treatment and medical support. Seizures make up about 1% of all emergency department visits for pediatric patients, and at least 5% of pediatric patients will have a seizure by the time they are 16 years old. Children younger than one year of age are commonly affected by new and unprovoked seizures.2 Seizures can result in continuous muscular activity, which leads to tissue breakdown because of anaerobic metabolism as well as decreasing oxygen and glucose to the brain causing brain ischemia and neuronal death. So, the seizures must be controlled rapidly to decrease the systemic as well as brain damage.3,4 First-line anticonvulsants for the treatment of acute seizures are benzodiazepines. Diazepam is frequently used for the treatment of seizures because it can be delivered either intravenously or rectally. It is lipophilic so does not have proper intramuscular absorption. Precious time is spent in getting intravenous access or per rectal catheterization. While midazolam, is a lipid-soluble benzodiazepine, rapidly absorbed after intramuscular (IM) injection.5,6 For managing seizure, the drug should be sufficiently potent to allow small volume and an administration that is quick, easy, and safe with quick action and little monitoring.7 Intramuscular midazolam meets these criteria and may be useful for the treatment of seizures, but more trials are needed to see the safety and efficacy of this therapy in the pediatric population.8 A major chunk of the seizures may occur out of the hospital. For the parents its frightening to see their kid in fits. Usually these parents immediately take their child to the nearby hospital or clinic. But it's not possible for all the parents, because in many areas health facilities are not present. Hence these patients are at increased risk for sustaining post ictal brain damage. There is a long-awaited wish that how to prevent this brain damage. A lot of options are tried nowadays and also in the past, like rectal diazepam, sublingual midazolam, but unfortunately most such options are not without risks.

The objective of this study was to compare the time taken by intramuscular midazolam to stop the seizure as compared to intravenous diazepam in emergency cases in the pediatric age group.

ELIGIBILITY:
Inclusion Criteria:

* Patients presented to the pediatric emergency, with all types of seizures, aged 3 months to 5 years.

Exclusion Criteria:

* 1. Children who already had intravenous access. 2. Children who had signs of clinical heart failure like tachycardia, tachypnea, and hepatomegaly.

  3. Children who had any severe systemic disease like renal disorder, liver disorder, and Beta Thalassemia major.

  4. Known allergy to midazolam or diazepam 5. Children who had hypoglycemia as the known cause of seizure 6. Children with other known causes of fits, like hypocalcemia, CKD, Hypoparathyroidism, Renal Tubular Acidosis

Ages: 3 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Fits Controlled | 300 seconds
  Treatment was considered successful if seizures stopped within 300 seconds of administering the drug. If seizures were not controlled within 300 seconds, Treatment failures were marked. other anticonvulsants were tried.

CONTACTS AND LOCATIONS:
Locations (1):
- Khyber Teaching Hospital, Peshawar, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hosseini F, Nikkhah A, Afkhami Goli M. Serum Zinc Level in Children with Febrile Seizure. Iran J Child Neurol. 2020 Winter;14(1):43-47. PMID 32021627
- [Background] Santillanes G, Luc Q. Emergency department management of seizures in pediatric patients. Pediatr Emerg Med Pract. 2015 Mar;12(3):1-25; quiz 26-7. PMID 25799698
- [Background] Scott RC. What are the effects of prolonged seizures in the brain? Epileptic Disord. 2014 Oct;16 Spec No 1(Spec No 1):S6-11. doi: 10.1684/epd.2014.0689. PMID 25323416
- [Background] Zilberter Y, Zilberter M. The vicious circle of hypometabolism in neurodegenerative diseases: Ways and mechanisms of metabolic correction. J Neurosci Res. 2017 Nov;95(11):2217-2235. doi: 10.1002/jnr.24064. Epub 2017 May 2. PMID 28463438
- [Background] Kienitz R, Kay L, Beuchat I, Gelhard S, von Brauchitsch S, Mann C, Lucaciu A, Schafer JH, Siebenbrodt K, Zollner JP, Schubert-Bast S, Rosenow F, Strzelczyk A, Willems LM. Benzodiazepines in the Management of Seizures and Status Epilepticus: A Review of Routes of Delivery, Pharmacokinetics, Efficacy, and Tolerability. CNS Drugs. 2022 Sep;36(9):951-975. doi: 10.1007/s40263-022-00940-2. Epub 2022 Aug 16. PMID 35971024
- [Background] Humphries LK, Eiland LS. Treatment of acute seizures: is intranasal midazolam a viable option? J Pediatr Pharmacol Ther. 2013 Apr;18(2):79-87. doi: 10.5863/1551-6776-18.2.79. PMID 23798902
- [Background] Agarwal SK, Cloyd JC. Development of benzodiazepines for out-of-hospital management of seizure emergencies. Neurol Clin Pract. 2015 Feb;5(1):80-85. doi: 10.1212/CPJ.0000000000000099. PMID 29443201
- [Background] Alansari K, Barkat M, Mohamed AH, Al Jawala SA, Othman SA. Intramuscular Versus Buccal Midazolam for Pediatric Seizures: A Randomized Double-Blinded Trial. Pediatr Neurol. 2020 Aug;109:28-34. doi: 10.1016/j.pediatrneurol.2020.03.011. Epub 2020 Mar 16. PMID 32387007